CLINICAL TRIAL: NCT00478621
Title: A Multicentre Study to Evaluate the Safety and Immunogenicity of GSK Biologicals' HPV Vaccine (GSK1674330A) in Healthy Female Subjects Aged 18-25 Years.
Brief Title: Human Papillomavirus Vaccine Safety & Immunogenicity Trial in Healthy Young Adult Women With HPV Vaccine (GSK1674330A)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 109836
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Infections, Papillomavirus
Keywords: HPV
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant

ARMS (6):
- Group A (Experimental)
  Interventions: Biological: GSK Biologicals' HPV vaccine (GSK1674330A)
- Group B (Experimental)
  Interventions: Biological: GSK Biologicals' HPV vaccine (GSK1674330A)
- Group C (Experimental)
  Interventions: Biological: GSK Biologicals' HPV vaccine (GSK1674330A)
- Group D (Experimental)
  Interventions: Biological: GSK Biologicals' HPV vaccine (GSK1674330A)
- Group E (Experimental)
  Interventions: Biological: GSK Biologicals' HPV vaccine (GSK1674330A)
- Group F (Active Comparator)
  Interventions: Biological: Cervarix TM

INTERVENTIONS:
Biological: GSK Biologicals' HPV vaccine (GSK1674330A) — Intramuscular administration, 5 different formulations
  Arms: Group A; Group B; Group C; Group D; Group E
Biological: Cervarix TM — Intramuscular administration
  Other Names: GSK Biologicals' HPV vaccine (580299)
  Arms: Group F

SUMMARY:
Infection with human papillomavirus (HPV) has been clearly established as the central cause of cervical cancer. Indeed, certain oncogenic types of HPV can infect the cervix (part of the uterus or womb). This infection may go away by itself, but if it does not go away (this is called persistent infection), it can lead in women over a long period of time to cancer of the cervix. GlaxoSmithKline Biologicals has developed a HPV vaccine against the oncogenic types HPV-16 and HPV-18 formulated with the AS04 adjuvant (control vaccine) and is also evaluating novel HPV vaccines formulations. This study will evaluate a novel GSK Biologicals' HPV vaccine (GSK1674330A) in terms of safety and immunogenicity compared to the control vaccine. There will be different levels of blinding in the study.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* A woman whom the investigator believes can and will comply with the requirements of the protocol.
* A woman between, and including, 18 and 25 years of age at the time of the first vaccination.
* Written informed consent must be obtained from the subject prior to enrolment.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Subject must be of non-childbearing potential, or if of child bearing potential, she must have a negative pregnancy test and she must be using adequate contraceptive precautions for 30 days prior to the first vaccination and must agree to continue such precautions for two months after completion of the vaccination series.
* Subject who has had no more than 6 lifetime sexual partners prior to enrolment.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use up to six months after last dose of vaccine.
* Concurrently participating in another clinical study, at any time during the study period (up to six months after last dose of vaccine), in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose or planned during the study period up to one month after last dose of vaccine.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before and 30 days after (i.e. days 0-29) the first dose of study vaccine. Planned administration/administration of routine vaccines up to 8 days before the first dose of study vaccine is allowed. Enrolment will be deferred until the subject is outside of specified window.
* Pregnant or breastfeeding. Women must be at least 3 months post-pregnancy and not breastfeeding to enter the study.
* A woman planning to become pregnant or planning to discontinue contraceptive precautions during the study period, up to two months after the last vaccine dose.
* Previous vaccination against HPV or planned administration of any HPV vaccine other than that foreseen by the study protocol during the study period.
* Previous administration of components of the investigational vaccine
* Any medically diagnosed or suspected immunodeficient condition based on medical history and physical examination of allergic disease, suspected allergy or reactions likely to be exacerbated by any component of the study vaccines.
* Hypersensitivity to latex.
* Known acute or chronic, clinically significant pulmonary, cardiovascular, neurologic, hepatic or renal functional abnormality, as determined by previous physical examination or laboratory tests.
* Cancer or autoimmune disease under treatment.
* History of allergic disease, suspected allergy or reactions likely to be exacerbated by any component of the study vaccines.
* History of having had colposcopy or has planned a colposcopy to evaluate an abnormal cervical cytology test.
* Received immunoglobulins and/or blood product within 3 months preceding enrolment or planned administration during the study period up to one month after the last dose of vaccine. Enrolment will be deferred until the subject is outside of specified window.
* Acute disease at the time of enrolment.
* Heavy bleeding (menstruation or other) or heavy vaginal discharge in which a cervical sample cannot be collected. Enrolment will be deferred until condition is resolved according to investigators medical judgement.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 540 (Actual)
Dates: Start 2007-05-25 (Actual); Primary Completion 2008-06-30 (Actual); Study Completion 2008-10-13 (Actual)

PRIMARY OUTCOMES:
Occurrence, intensity and relationship to vaccination of any solicited local or general symptoms | Within 7 days after each vaccine dose

SECONDARY OUTCOMES:
Occurrence of serious adverse events | Up to one month after the last dose of vaccine
Occurrence, intensity and relationship to vaccination of any unsolicited symptom | Within 30 days after each vaccine dose
Occurrence of clinically relevant abnormalities in biochemical and hematological parameters | Assessed at Month 0, one month and six months after the last dose of vaccine
Occurrence of serious adverse events during the extended safety follow-up | Up to six months after the last dose of vaccine
Occurrence of pregnancy and pregnancy outcomes, new onset chronic diseases or medically significant conditions, regardless of causal relationship to vaccination | Throughout the study period (Month 0 up to six months after the last dose of vaccine)
HPV-16 and HPV-18 seropositivity rates and GMTs before the second dose of vaccine | One month after the second dose of vaccine, and six months after the last dose of vaccine
Seropositivity rates to other defined HPV types and GMTs before the second dose of vaccine | One month after the second dose of vaccine and at one month and six months after the last dose of vaccine
HPV-16 and -18 seropositivity rates and GMTs | One month after the last dose of vaccine

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Belgium (3):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Wilrijk

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Van Damme P, Leroux-Roels G, Simon P, Foidart JM, Donders G, Hoppenbrouwers K, Levin M, Tibaldi F, Poncelet S, Moris P, Dessy F, Giannini SL, Descamps D, Dubin G. Effects of varying antigens and adjuvant systems on the immunogenicity and safety of investigational tetravalent human oncogenic papillomavirus vaccines: results from two randomized trials. Vaccine. 2014 Jun 17;32(29):3694-705. doi: 10.1016/j.vaccine.2014.03.040. Epub 2014 Mar 25. PMID 24674663
- See also: Results for study 109836 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/109836?search=study&b''#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 109836 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109836 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109836 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109836 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109836 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 109836 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register